CLINICAL TRIAL: NCT07040683
Title: Negative Pressure Wound Therapy for Split Thickness Skin Grafting to the Lower Leg After Excision of Skin Tumour: The Legs Trial - A Multicentre Randomised Study
Brief Title: Negative Pressure Wound Therapy for Split Thickness Skin Grafting to the Lower Leg After Excision of Skin Tumour: A Multicentre Randomised Study
Acronym: LEGS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Pooya Rajabaleyan, Negative pressure wound therapy for split thickness skin grafting to the lower leg after excision of skin tumour: The Legs Trial - A multicentre randomised study, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-05592-01
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Skin Transplantation; Skin Grafting; Split Thickness Skin Graft; Negative-Pressure Wound Therapy; Postoperative Complications; Surgical Wound Infection; Lower Extremity; Skin Cancer; Skin Tumour; Wound Healing; Bandages; Leg
Keywords: Skin Transplantation; Skin Grafting; Split Thickness; Negative-Pressure Wound Therapy; Postoperative Complications; Surgical Wound Infection; Lower Extremity; Wound Healing; Bandages; Leg; Skin Neoplasms; Skin Cancer
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection; Skin Neoplasms | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either negative pressure wound therapy (NPWT) or traditional dressings after split-thickness skin grafting to the lower leg. Each participant will remain in their assigned treatment group for the duration of the study, with outcomes assessed at follow-up visits and by medical record review up to three months postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy (NPWT) (Experimental): Participants in this arm will receive negative pressure wound therapy (NPWT) applied over the split-thickness skin graft after excision of a skin tumour on the lower leg. NPWT will be applied according to manufacturer instructions, using a protective interface layer and continuous negative pressure of -125 mmHg until postoperative day 5.
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)
- Traditional Dressings (Active Comparator): Participants in this arm will receive traditional dressings applied over the split-thickness skin graft after excision of a skin tumour on the lower leg. The dressing will include a protective silicone interface layer and foam dressing with gentle compression, left undisturbed until postoperative day 5.
  Interventions: Other: Traditional Dressing

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (NPWT) — Negative pressure wound therapy (NPWT) applied over the split-thickness skin graft on the lower leg after tumour excision. A protective silicone interface layer will be used, with continuous negative pressure of -125 mmHg applied until postoperative day 5, unless earlier change is clinically indicated.
  Other Names: VAC Therapy; Negative Pressure Dressing
  Arms: Negative Pressure Wound Therapy (NPWT)
Other: Traditional Dressing — Traditional dressing applied over the split-thickness skin graft on the lower leg after tumour excision. The dressing consists of one or more layers of foam dressing applied on top, which may or may not be fixed with sutures according to surgeon preference, and an elastic bandage applied over the foam to provide gentle, even compression and immobilisation of the graft. The dressing will remain undisturbed until postoperative day 5 unless earlier change is clinically indicated.
  Arms: Traditional Dressings

SUMMARY:
The goal of this clinical trial is to compare the effect of negative pressure wound therapy (NPWT) versus traditional dressings on the incidence of transplant infection in adult patients undergoing split-thickness skin grafting (STSG) to the lower leg following excision of a skin tumour. The main questions it aims to answer are:

Does NPWT reduce the incidence of transplant infection within three months after STSG?

Does NPWT improve secondary outcomes such as graft take, reduce reoperations, complications, and resource use?

Researchers will compare patients treated with NPWT to patients treated with traditional dressings to see if NPWT results in lower infection rates and better clinical outcomes.

Participants will:

Undergo excision of a skin tumour on the lower leg followed by STSG.

Be randomized to receive either NPWT or traditional dressings applied over the graft.

Follow a structured postoperative care and mobilisation schedule.

Attend follow-up visits at day 5 and day 14 postoperatively and be monitored through medical record review up to three months after surgery.

DETAILED DESCRIPTION:
Split-thickness skin grafting (STSG) to the lower leg is a common surgical procedure performed after excision of skin tumours, particularly when primary closure is not feasible. Although the technique is well established, postoperative infections and graft-related complications remain a clinical challenge, especially in lower leg wounds, which are prone to oedema and mechanical stress.

Negative pressure wound therapy (NPWT) has been introduced as an alternative to traditional dressings for skin grafts. NPWT applies controlled suction to the wound environment, promoting fluid removal, enhancing blood flow, and potentially improving graft adherence and reducing infection risk. However, current evidence for NPWT in lower leg grafting is limited and inconclusive.

The Legs Trial is a multicentre, randomised controlled trial designed to compare NPWT with traditional dressings in adult patients undergoing STSG to the lower leg after tumour excision. The primary objective is to assess whether NPWT reduces the incidence of transplant infections within three months. Secondary outcomes include graft loss, reoperations, postoperative complications, hospital stay, and healthcare resource use.

Patients will be randomised to receive either NPWT or traditional dressing at the time of surgery. All patients will follow a structured postoperative mobilisation protocol and attend follow-up visits for outcome assessment.

The trial aims to generate high-quality evidence to inform best practices in postoperative management of lower leg skin grafts and optimise patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Undergoing excision of a skin tumour on the lower leg with planned coverage using split-thickness skin grafting (STSG)
* Eligible procedures include primary excision, secondary excision, or extended excision performed at the same site as a previous tumour surgery
* Ability to provide written informed consent
* Ability to comply with postoperative instructions and follow-up visits

Exclusion Criteria:

* Inability to follow postoperative instructions due to cognitive impairment, dementia, or significant language barriers
* Inability to provide informed consent
* Severe systemic illness, including:
* Ongoing sepsis
* Advanced heart failure
* End-stage renal or liver disease
* Active chemotherapy within the previous three months
* Ongoing treatment with immunosuppressive medications, including:
* Systemic corticosteroids (e.g., prednisone >20 mg/day or equivalent)
* Calcineurin inhibitors (e.g., cyclosporine, tacrolimus)
* Antimetabolites (e.g., methotrexate, azathioprine, mycophenolate mofetil)
* mTOR inhibitors (e.g., sirolimus, everolimus)
* Biologic therapies (e.g., rituximab, TNF inhibitors, IL-6 inhibitors, IL-1, IL-17, IL-23 inhibitors)
* Targeted molecular therapies (e.g., JAK inhibitors such as tofacitinib, baricitinib)
* Other immunosuppressive drugs
* Previous radiation therapy to the surgical site
* Presence of severe skin disease affecting the planned graft recipient site (e.g., advanced psoriasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of transplant infection within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  Transplant infection defined as clinical infection of the skin graft diagnosed by a physician or confirmed by microbiological culture, occurring within 3 months after initial tumor excision and split-thickness skin grafting to the lower leg.

SECONDARY OUTCOMES:
Graft loss within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  Graft loss defined as <90% graft take at the graft site within 3 months after index surgery.
Reoperation within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  Proportion of participants requiring reoperation related to the graft site within 3 months after index surgery.
Bleeding within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  Incidence of clinically significant bleeding at the graft site requiring medical intervention within 3 months after index surgery.
Systemic complications within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  Incidence of systemic complications including deep vein thrombosis, pulmonary embolism, or myocardial infarction occurring within 3 months after index surgery.
Mortality within 3 months after index surgery | From date of index surgery until 3 months postoperatively.
  All-cause mortality within 3 months after index surgery.
Length of hospital stay | From date of index surgery until 3 months postoperatively.
  Number of inpatient days related to the graft procedure.
Healthcare resource use within 3 months | From date of index surgery until 3 months postoperatively.
  Healthcare resource use based on costs of NPWT, traditional bandages, number of outpatient visits, use of antibiotics, and total days of hospitalisation within 3 months after index surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Plastic and Reconstructive Surgery and Dept. of Health Sciences, Skåne University Hospital, Malmö, Sweden., Malmo, Sweden